CLINICAL TRIAL: NCT05917431
Title: Phase 2 Study of Stereotactic Body Radiation Therapy Plus Tislelizumab and Regorafenib in Unresectable or Oligometastatic Hepatocellular Carcinoma
Brief Title: Phase 2 Study of SBRT Plus Tislelizumab and Regorafenib in Unresectable or Oligometastatic HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wang weihu, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-LiCaS2
Record Dates: First submitted 2023-05-24; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Unresectable Hepatocellular Carcinoma; Oligometastatic Disease
MeSH Terms: interventions — Radiosurgery; tislelizumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT plus Tislelizumab and Regorafenib (Experimental): Participants will receive SBRT (8 Gy × 3-5 fractions) to all visible lesions. Systemic treatment (tislelizumab and regorafenib) will start concurrently and last for 2 years, or until disease progression, intolerable side-effects or death. Tislelizumab will be delivered every 21 days at a dose of 200mg, and regorafenib will be given at a dose of 120mg for the first 21 days of a 28-day cycle. Appropriate dose adjustments of regorafenib will be made if side-effects are intolerable, while the dose of tislelizumab should not be adjusted, but could be paused.
  Interventions: Combination Product: SBRT plus tislelizumab and regorafenib

INTERVENTIONS:
Combination Product: SBRT plus tislelizumab and regorafenib — Participants will receive SBRT plus tislelizumab and regorafenib concurrently

SUMMARY:
The goal of this phase 2 prospective clinical trial is to learn about the efficacy and safety of stereotactic body radiation therapy (SBRT) plus immunotherapy and targeted therapy in patients with unresectable or oligometastatic hepatocellular carcinoma (HCC).

The main question to answer is: Whether combing SBRT with immunotherapy and targeted therapy could prolong PFS. Participants will receive SBRT to all visible lesions and concurrent systemic immunotherapy and targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Eastern Cooperative Oncology Group performance status of 0-1
* clinical or pathological diagnosis of HCC
* with unresectable locally advanced or oligometastatic HCC (metastatic lesions ≤ 5, metastatic organs ≤ 3, may involve extrahepatic lymph nodes or distant organs apart from brain)
* at least one measurable lesion according to mRECIST criteria
* all lesions could be included in radiation target volume
* Child-Pugh A or B (7 scores) liver function
* patients are allowed to receive systemic therapy previously other than tislelizumab plus regorafenib
* adequate hematological and renal function
* life expectancy ≥ 3 months；
* willing to participate in the study and give written informed consent

Exclusion Criteria:

* a history of liver transplantation
* with severe cirrhosis complications, including a history of esophagogastric variceal bleeding, hepatic encephalopathy, and massive ascites
* with active autoimmune diseases or a history of autoimmune disease
* with human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
* allergic to the ingredient of tislelizumab or regorafenib
* with recurrent lesions treated with radiotherapy previously
* prescribed radiation does could not be delivered due to dose limits to organs at risk (OAR)
* intolerable to radiation or systemic treatment because of cardiac insufficiency, uncontrolled high blood pressure
* a history of other malignancies, except cured basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | From the date of treatment beginning until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Progression-free survival

SECONDARY OUTCOMES:
OS | From the date of treatment beginning until the date of death from any cause, assessed up to 48 months
  Overall survival
Recurrence pattern | From the date of treatment beginning until the date of last follow-up, assessed up to 48 months
  Number of participants with recurrence, which will be classified according to site of recurrence (specific organs), time interval between treatment beginning and recurrence, the relationship with the area of irradiation (in-field/out field), and whether new lesion(s) according to mRECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No